CLINICAL TRIAL: NCT05859022
Title: Comparison of Metabolic Effects of Bariatric Arterial Embolization vs. Bariatric Surgery
Brief Title: Metabolic Effects of Bariatric Arterial Embolization vs Bariatric Surgery
Acronym: BEOD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Nova de Lisboa (Other)
Collaborators: cruz vermelha hospital (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BEOD trial
Record Dates: First submitted 2023-04-03; First posted 2023-05-15 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Obesity; Type2diabetes; Bariatric Surgery Candidate; Metabolic Disease
Keywords: bariatric surgery; embolization; intensive medical therapy; BMI; glycemia
MeSH Terms: conditions — Obesity; Metabolic Diseases | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: Patients assigned for one of 2 arms: Roux-en-Y gastric By-pass (RYGB),bariatric arterial embolization (BAE).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Roux-en-Y gastric By-pass (RYGB) (Experimental): RYGB procedure requires 1-2 hours of operating time and two to three days length of hospital stay. Use the Kit-RYGB by J& company.
  Interventions: Other: Roux-en-Y gastric By-pass (RYGB) surgery
- Bariatric Arterial Embolization (BAE) (Experimental): Embosphere Microspheres (EM) are designed to offer controlled, target embolization. BAE procedure requires 1hour of operating time and one day length of hospital stay. Use the Kit by Merit MedicalCompany.
  Interventions: Other: Bariatric Arterial Embolization (BAE) procedure

INTERVENTIONS:
Other: Roux-en-Y gastric By-pass (RYGB) surgery — RYGB procedure requires 1-2 hours of operating time and two to three days length of hospital stay. Use the Kit-RYGB by J& company.
  Arms: Roux-en-Y gastric By-pass (RYGB)
Other: Bariatric Arterial Embolization (BAE) procedure — use of Embosphere Microspheres (EM) that are designed to offer controlled, target embolization.
  Arms: Bariatric Arterial Embolization (BAE)

SUMMARY:
Obesity and Type 2 diabetes mellitus (DMT2) are two of the most common chronic diseases of the Western society. Obesity is one critical factor in DMT2 development, with weight loss having profound beneficial effects on DMT2 and improving the metabolic pathophysiology leading to hyperglycemia.

Observational studies reported that surgical intervention of morbid obesity achieved significant improvement of resolution of DMT2, both in short and long-term. Bariatric surgery has been considered the best option for treatment of diabetic obese patients, with the laparoscopic Roux-en-Y Gastric Bypass being the gold standard of the surgical treatment. Bariatric arterial embolization (BAE) technique has proved to be safe effective for weight loss in obese patients, but its metabolic effects have not been studied yet. The hypothesis of the study is that BAE is effective for the resolution of DMT2 inpatients with BMI between 30-43 Kg/m2. The aim is to assess DMT2 remission after BAE and bariatric surgery, to analyze potential conditioning factors, and to compare remission criteria between bariatric surgery and BAE.

DETAILED DESCRIPTION:
The present project is a prospective, randomized, no-blinded, controlled and interventional clinical single- center study, which seeks to compare the impact of the following interventions: Roux-en-Y gastric By-pass (RYGB) and bariatric arterial embolization (BAE) on metabolic control in patients with DMT2 and BMI between 30-43 Kg/m2 over 2 years.

Study initial recruitment will be achieved by an awareness campaign, which will emphasize a study of methods of diabetes management and include identification of patients into treatment at Cruz Vermelha Hospital. The investigator will initially pre-screen patients for the inclusion and exclusion criteria. Detailed information regarding of Diabetes, Obesity and randomization arms of the study would be provided in service meeting.

Evaluation of the inclusion and exclusion criteria will occur both at the initial screening visit and the baseline visit prior to randomization. Patients who fail to be include during initial screening may be considered for re-consenting when clinically appropriate, and will have screening/baseline procedures repeated at the discretion of the Investigator. Patients who fail to be include during initial screening based on glycated hemoglobin (HbA1c) and or BMI and are re/screened within 6 months, will only have the baseline HbA1c and BMI repeated.

On visit 2 (after 30 days) the 60 patients randomized per study arm for embolization or surgery procedures will be evaluated by the anaesthetist. RYGB or BAE will be scheduled as soon as possible after randomization.

After BAE or surgery, patients will be followed 1, 3, 6 and 12 months. At 12 months visit patients will be evaluated for primary endpoint of percent of treatment group achieving HbA1c ≤ 6%.

Pre-specified secondary outcomes include measures of glycaemic control, weight loss, mean blood pressure, lipid levels, renal function, assessment of diabetes quality of life (DQoL) and biomarkers in blood. Also, metabolic parameters and other markers will be evaluated from liver and adipose tissue biopsies collected at the beginning of the RYGB surgery to correlate with biochemical evaluations.

During the follow-up visits primary and secondary outcomes will be evaluated by different techniques and approaches: body weight loss will be evaluated by bioimpedance analysis; blood will be collected for HbAlc, fasting glucose, lipids, comprehensive Metabolic Panel, Urinalysis (microalbumin and creatinine) and hepatogram by common clinical analysis; the diabetes quality of life (DQoL) question; liver and adipose tissues will be collected during the surgical procedure to asses by western blot the levels of each adenosine receptors, adipokynes, cytokines and inflammatory markers receptors.

ELIGIBILITY:
Inclusion Criteria:

* criteria:

  1. Is the candidate for general anesthesia.
  2. Body Mass Index (BMI) between 33 and 43 Kg/m2
  3. Patients have a biochemical evidence of Type 2 Diabetes Mellitus (DMT2) confirmed by American Diabetes Association (ADA) criteria:

     3.1) treated - HbA1c 7,1%; 3.2) If untreated- fasting 2-hour plasma glucose level of 200 mg/dL during an oral glucose tolerance test and a HbA1c of 7,1%.
  4. Willing, able, and mentally competent to provide written informed consent.
  5. Able o understand the options and to comply with the requirements of each program.
  6. Have a negative urine pregnancy test at screening and baseline visits (prior surgery and Embolization) for women of childbearing potential.
  7. Female patients must agree to use reliable method of contraception for 2 years.

Exclusion Criteria:

1. Prior bariatric surgery of any kind.
2. Prior complex abdominal surgery including splenectomy, upper GI, anti-reflux surgery and trauma.
3. Abdominal, thoracic, pelvic and/or obstetric-gynaecologic surgery within 3 months or at the discretion of the surgery.
4. Cardiovascular conditions including uncompensated congestive heart failure, dysrhythmia, history of stroke, or uncontrolled hypertension (defined as medically treated with the mean of 3 separate measurements systolic blood pressure (SBP)> 180 mmHg or diastolic blood pressure (DBP) >110mmHg). Patients with coronary artery disease (CAD) that have been successfully treated with coronary artery by-pass graft (CABG) or percutaneous coronary intervention (PCI) or are 1 year after implantation of drug eluting stent and have no evidence of active ischemia are eligible.
5. Known history of chronic liver disease (except for NAFLD/NASH), hepatitis, positive serologic test result for hepatitis B surface antigen and/or hepatitis C antibody, alpha-1-antitrypsin deficiency.
6. Gastrointestinal disorders including a known history of celiac disease and/or other malabsorptive disorders or inflammatory bowel disease (Chron's disease or ulcerative colitis).
7. Psychiatric disorders including dementia, active psychosis, severe depression requiring >2 medications, history of suicide attempts, alcohol or drugs abuse with previous 12months.
8. Pregnancy.
9. Malignancy within 5 years (except squamous cell and basal cell cancer of skin).
10. Anaemia defined as haemoglobin less than 9 in females and 10 in males.
11. Any medical condition requiring anticoagulation therapy that cannot be temporarily discontinued for surgical or embolic approach.
12. Any condition or major illness that, in the investigator's judgment, places the subject at undue risk by participating in the study.
13. Use of investigational therapy or participation in any other clinical trial within 12 weeks prior to signing the informed consent form.
14. Severe pulmonary disease.
15. American Society of Anesthesiologists (ASA) physical status class IV or higher.
16. History of allergy to iodinated contrast media

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-06-16 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Number of participants with glycated haemoglobin < 6% | 12 months
  The primary outcome of the study will be a level of glycated haemoglobin of 6.0% or less without the use of diabetes medications.

SECONDARY OUTCOMES:
Determination of glycemic level (mg/dL) | up to 48 months
  Measures of glycemic control by evaluating glycemic level at fast in the blood in mg/dL. less than 126mg/dL will represent a good glycemic control
Weight evaluation in Kg | up to 48 months
  Evaluation of weight loss in Kg from the first appointment and during the different admissions time-points of each patient
Blood pressure measurement | up to 48 months
  Evaluation of mean blood pressure in mmHg in the first appointment and during the entire trial
Determination of lipid levels | up to 48 months
  Evaluation of lipid levels in the first appointment and during the entire trial
Determination of renal function | up to 48 months
  Evaluation of renal function by measuring creatinine levels in the blood in the first appointment and during the entire trial
Assess diabetes quality of life (DQoL) questionnaire | up to 48 months
  Evaluation of diabetes quality of life (DQoL) questionnaire in the first appointment and during the entire trial. it will measure reliability and validity of a diabetes quality-of-life and will measure the diabetes control and complications. The instrument provides an overall scale score ranging from 0 (lowest DQoL score) to 100 (highest DQoL score), as well as four subscale scores for: 1- satisfaction with treatment, 2- impact of treatment, 3- worry about the future effects of diabetes, and 4- worry about social/vocational issues.
Evaluation of adenosine metabolism in liver and adipose tissue biopsies | At the beginning of the RYGB surgery
  evaluation of adenosine receptors protein levels (A1R, A2aR, A2bR) (given in % of protein levels from control) on liver and adipose tissue collected at the beginning of RYGB surgery. the evaluation of the 3 receptors levels will allow to evaluate adenosine metabolism in a whole.
Evaluation of adipokines in adipose tissue biopsies | At the beginning of the RYGB surgery
  Evaluation of adipokines protein levels (leptin, adiponectin and resistin; given in % of protein levels from control) on adipose tissue collected at the beginning of RYGB surgery. the evaluation of the adipokines levels will allow to evaluate overall adipose tissue function.
Evaluation of cytokines in liver and adipose tissue biopsies | At the beginning of the RYGB surgery
  evaluation of cytokines protein levels [interleukin 10 (IL10), tumor necrosis factor alpha (TNFalpha), interleukin 6 (IL6); given in % protein levels from the control) on liver and adipose tissue collected at the beginning of RYGB surgery. the evaluation of cytokines on both tissues will allow to determine the overall inflammatory status of the tissues.
Evaluation of inflammatory receptors levels in liver and adipose tissue biopsies | At the beginning of the RYGB surgery
  evaluation of inflammatory receptors protein levels (IL10 receptor, TNFalpha receptor, IL6 receptor; given in % protein levels from the control) on liver and adipose tissue collected at the beginning of RYGB surgery. the evaluation of cytokines on both tissues will allow to determine the overall inflammatory status of the tissues.

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo O. Oliveira, MD, Principal Investigator — cruz vermelha hospital
Locations (1):
- Cruz Vermelha Hospital, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: Yes
all individual participant data (IPD) that underlie results in publications and a Philosophy doctor (PhD) thesis
Supporting Information: Study Protocol, SAP, CSR
Time Frame: From 24months some data will be shared and till the end of the project at 48months after recruitment of all patients
Access Criteria: Results from the present study will be presented in several national and international meetings and published in scientific journals. The PhD dissertation will be done by compiling the articles published in the context of this project.